CLINICAL TRIAL: NCT01922102
Title: A 12-month, Phase III, Randomized, Double-masked, Multicenter, Active-controlled Study to Evaluate the Efficacy and Safety of Two Individualized Regimens of 0.5mg Ranibizumab vs. Verteporfin PDT in Patients With Visual Impairment Due to Choroidal Neovascularization Secondary to Pathologic Myopia
Brief Title: Efficacy and Safety of Ranibizumab 0.5 vs Verteporfin PDT in Patients With Visual Impairment Due to Choroidal Neovascularization Secondary to Pathologic Myopia
Acronym: Brilliance
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRFB002F2302
Record Dates: First submitted 2013-08-12; First posted 2013-08-14 (Estimated); Results first posted 2019-06-24 (Actual); Last update posted 2019-06-24 (Actual); Status verified 2019-03

CONDITIONS: Visual Impairment Due to Choroidal Neovascularization (CNV) Secondary to Pathologic Myopia (PM)
Keywords: vision loss,PM,CNV,ranibizumab,verteporfinPDT,Brilliance
MeSH Terms: conditions — Choroidal Neovascularization | interventions — Ranibizumab; Verteporfin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (Experimental): 0.5 mg ranibizumab driven by visual acuity stability criteria
  Interventions: Drug: Ranibizumab 0.5mg
- Group II (Experimental): 0.5 mg ranibizumab driven by disease activity criteria
  Interventions: Drug: Ranibizumab 0.5 mg
- Group III (Active Comparator): verteporfin PDT
  Interventions: Drug: Verteporfin PDT

INTERVENTIONS:
Drug: Ranibizumab 0.5mg — 0.5 mg ranibizumab (intravitreal injections)
  Other Names: Lucentis
  Arms: Group I
Drug: Ranibizumab 0.5 mg — 0.5 mg ranibizumab (intravitreal injections)
  Other Names: Lucentis
  Arms: Group II
Drug: Verteporfin PDT — Verteporfin for intravenous injection delivered by intravenous infusion followed by the light application
  Other Names: Visudyne
  Arms: Group III

SUMMARY:
This study was designed to evaluate the efficacy and safety of two different dosing regimens of 0.5 mg ranibizumab given as intravitreal injection in comparison to verteporfin PDT in patients with visual impairment due to choroidal neovascularization secondary to pathologic myopia (PM)

DETAILED DESCRIPTION:
This was a phase III, multi-center, randomized, double-masked, active-controlled study comparing 0.5 mg ranibizumab vs. vPDT therapy. The study included 15 scheduled visits over 12 months, and there were to be two additional visits (2a, 3a) for subset of patients in whom PK analysis were performed.

There were 3 periods in this study: Screening period-from Day -14 to Baseline; Treatment period-from Baseline to Month 11; Follow-up period-from Month 11 to Month 12 Patients entered the 11 months Treatment period at Visit 2 (Day 1) if eligibility criteria were met and were randomized in three treatment groups Group I ranibizumab 0.5 mg driven by VA stability criteria or Group II ranibizumab 0.5 mg driven by disease activity criteria or Group III vPDT (randomization ratio of 2:2:1) and received first treatment of either a ranibizumab injection and sham vPDT or sham injection and active vPDT and will return to the clinical center within 7 days to undergo safety assessments as well as assessments of the effect of treatment by the evaluating investigator. The following visits were performed at one month intervals starting at Visit 4 and continuing through Visit 14. At all monthly visits (at/from Month 2 for group I, at/from Month 1 for group II and at/from Month 3 for group III) the decision for treatment were made by the evaluating investigator based on the VA stability criteria and on the disease activity criteria. At Month 3 (visit 6) and at all following monthly visits for all three groups one of the three options can recommended by evaluating investigator: a) ranibizumab 0.5 mg, b) ranibizumab 0.5 mg + vPDT; c) vPDT. The treating investigator were then perform treatment based on randomization and masking requirements.

At each monthly visit, patients had a safety evaluation by the evaluating investigator prior to study treatment, consisting of visual acuity measurements, ophthalmic examinations and evaluation of adverse events and vital signs. Routine hematology, chemistry, and urinalysis profiles were obtained at Visit 6, 9 and 12 (Month 3, 6 and 9). At Month 12 several procedures and assessments were performed which are required at study completion visit.

ELIGIBILITY:
Inclusion Criteria:

* Visual impairment due to CNV secondary to PM.
* Best corrected visual acuity in the study eye > 24 and < 78 ETDRS letters.
* High myopia (> -6D),
* anterio-posterior elongation > 26 mm; posterior changes compatible with the pathologic myopia.
* Either CNV locations in the study eye: subfoveal, juxtafoveal, extrafoveal.

Exclusion Criteria:

* Some preexisting eye disorders or systemic diseases;-Blood pressure > 150/90 mmHg
* Prior focal/grid laser to the macular area -History of treatment with any anti-VEGF or verteporfin PDT in the study eye
* Intravitreal treatment with corticosteroids or intraocular surgery within last 3 months in the study eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 457 (Actual)
Dates: Start 2013-09-11 (Actual); Primary Completion 2016-09-14 (Actual); Study Completion 2016-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (35):
- China (18):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Chongqing, Chongqing Municipality
  - Novartis Investigative Site, Shantou, Guangdong
  - Novartis Investigative Site, Harbin, Heilongjiang
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Wuxi, Jiangsu
  - Novartis Investigative Site, Nanchang, Jiangxi
  - Novartis Investigative Site, Qingdao, Shandong
  - Novartis Investigative Site, Xi’an, Shanxi
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Tianjin, Tianjin Municipality
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Wenzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Chongqing
  - Novartis Investigative Site, Shanghai
- Novartis Investigative Site, Hong Kong, Hong Kong
- India (9):
  - Novartis Investigative Site, Chandīgarh, Haryana
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, Vanchiyoor, Kerala
  - Novartis Investigative Site, Bhubaneswar, Odisha
  - Novartis Investigative Site, Chennai, Tamil Nadu
  - Novartis Investigative Site, Coimbatore, Tamil Nadu
  - Novartis Investigative Site, Hyderabad, Telangana
  - Novartis Investigative Site, Angamaly
  - Novartis Investigative Site, New Delhi
- Novartis Investigative Site, Manila, National Capital Region, Philippines
- South Korea (2):
  - Novartis Investigative Site, Pusan
  - Novartis Investigative Site, Seoul
- Thailand (4):
  - Novartis Investigative Site, Khon Kaen, THA
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai
  - Novartis Investigative Site, Nakornphathom

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Randomized Set: consisted of all randomized patients. Patients were considered randomized when they had been given a randomization number.
Pre-assignment Details: In total, 457 patients were randomized into this study in a ratio of 2:2:1: 182 to Group I, 184 to Group II, and 91 to Group III.
Groups:
- Group III: verteporfin PDT (driven by disease activity). Patients received vPDT on Day 1. From Month 3, based on disease activity vPDT, Ranibizumab 0.5 mg, or combo of Ranibizumab and vPDT was selected for treatment
Period: Overall Study
Arm/Group | Group I | Group II | Group III
Started | 182 | 184 | 91
Completed | 173 | 175 | 83
Not Completed | 9 | 9 | 8
Not completed — Withdrawal by Subject | 7 | 3 | 7
Not completed — Physician Decision | 0 | 2 | 1
Not completed — Adverse Event | 1 | 2 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Administrative problems | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Randomized Set: consisted of all randomized patients. Patients were considered randomized when they had been given a randomization number.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I | Group II | Group III | Total
Number analyzed (Participants) | 182 | 184 | 91 | 457
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.0 (12.01) | 51.5 (12.13) | 49.1 (14.81) | 51.2 (12.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128 | 116 | 67 | 311
  Male | 54 | 68 | 24 | 146

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline BCVA to the Average Level of BCVA Over All Monthly Assessments From Month 1 to Month 3
Description: Best corrected visual acuity (BCVA) was tested using the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity (VA) charts testing protocol. VA measurements were taken in a sitting position at an initial test distance of 4 meters using ETDRS charts. The overall BCVA score was calculated using the BCVA worksheet, which was kept in the source data and the score was recorded in the eCRF.
Time Frame: From Baseline to Month 3
Population: Full Analysis Set (FAS): consisted of all patients to whom study treatment were assigned. Following the intent-to-treat principle, patients were analyzed according to the treatment group they were assigned to at randomization.
Measure: Mean (Standard Deviation); unit: ETDRS letters
Arm/Group | Group I | Group II | Group III
Number analyzed (Participants) | 182 | 184 | 91
ETDRS letters
  Baseline: number analyzed (Participants) | 181 | 184 | 89
  Baseline | 53.7 (12.65) | 54.2 (13.01) | 52.6 (12.29)
  Average Month 1 to Month 3 | 63.1 (12.80) | 63.9 (13.28) | 57.1 (13.21)
Statistical Analysis 1: Comparison: Group I vs Group III; 2 one-sided hypotheses were tested under the Type I error rate of 0.025, using the Hochberg procedure: H01: μRanibizumab-I - μvPDT ≤ 0 vs. HA1: μRanibizumab-I - μvPDT > 0 and H02: μRanibizumab-II - μvPDT ≤ 0 vs. HA2: μRanibizumab-II - μvPDT > 0, where μRanibizumab-I, μRanibizumab-II and μvPDT were the means of the primary efficacy variable for ranibizumab treatment Group I, ranibizumab treatment Group II, and vPDT treatment Group III, respectively; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Superiority could be claimed if the corresponding one-sided p-value was ≤ 0.025/2 = 0.0125, or if both one-sided p-values were ≤ 0.025; Mean Difference (Net) = 5.2, 95% CI 2-sided [3.3 to 7.1] — Differences in LS means and the two-sided 95% CIs are estimated from pairwise ANOVA (stratified) model
Statistical Analysis 2: Comparison: Group II vs Group III; The following 2 one-sided hypotheses were tested under the Type I error rate of 0.025, using the Hochberg procedure: H01: μRanibizumab-I - μvPDT ≤ 0 vs. HA1: μRanibizumab-I - μvPDT > 0 and H02: μRanibizumab-II - μvPDT ≤ 0 vs. HA2: μRanibizumab-II - μvPDT > 0, where μRanibizumab-I, μRanibizumab-II and μvPDT were the means of the primary efficacy variable for ranibizumab treatment Group I, ranibizumab treatment Group II, and vPDT treatment Group III, respectively; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 5.6, 95% CI 2-sided [3.5 to 7.6] — Differences in LS means and the two-sided 95% CIs are estimated from pairwise ANOVA (stratified) model

2. Secondary Outcome: Change From Baseline BCVA to the Average Level of BCVA Over All Monthly Assessments From Month 1 to Month 6
Description: Best corrected visual acuity (BCVA) was tested using the early treatment diabetic retinopathy study (ETDRS) VA testing protocol. VA measurements were taken in a sitting position at an initial test distance of 4 meters using ETDRS charts. The overall BCVA score was calculated using the BCVA worksheet, which was kept in the source data and the score was recorded in the eCRF.
  Between treatment comparison of 0.5 mg ranibizumab intravitreal injections driven by disease activity re-treatment criteria (Group II) versus 0.5 mg ranibizumab intravitreal injections driven by visual acuity stability criteria (Group I) based on the average BCVA change from Baseline to Month 1 through Month 6.
Time Frame: From Baseline to Month 6
Population: Full Analysis Set (FAS): Following the intent-to-treat principle, patients were analyzed according to the treatment group they were assigned to at randomization.
  FAS, modified last observation carried forward (LOCF), for comparison between ranibizumab treatment groups.): consisted of all patients to whom study treatment were assigned.
Measure: Mean (Standard Deviation); unit: ETDRS letters
Arm/Group | Group I | Group II | Group III
Number analyzed (Participants) | 182 | 184 | 91
ETDRS letters
  Baseline: number analyzed (Participants) | 182 | 184 | 89
  Baseline | 53.7 (12.65) | 54.2 (13.01) | 52.6 (12.29)
  Average Month 1 to Month 6: number analyzed (Participants) | 182 | 184 | 89
  Average Month 1 to Month 6 | 64.1 (12.77) | 64.9 (13.14) | 59.6 (12.99)
Statistical Analysis 1: Comparison: Group I vs Group II; Test type: Non-Inferiority or Equivalence — one-sided hypotheses were tested under the Type I error rate of 0.025, if H01 and H02 were rejected: H03: μRanibizumab-II - μRanibizumab-I ≤ -5 vs. HA3: μRanibizumab-II - μRanibizumab-I > -5. Otherwise, H03 was not to be considered as rejected; p < 0.001, Cochran-Mantel-Haenszel — Non-inferiority could be claimed if the corresponding one-sided p-value was ≤ 0.025; Mean Difference (Net) = 0.4, 95% CI 2-sided [-1.3 to 2.1] — Differences in LS means and the two-sided 95% CIs are estimated from pairwise ANOVA (stratified) model

3. Secondary Outcome: The Average Change in BCVA Score From Baseline to Month 1 Through Month 12
Description: Best corrected visual acuity (BCVA) was tested using the ETDRS VA testing protocol. VA measurements were taken in a sitting position at an initial test distance of 4 meters using ETDRS charts. The overall BCVA score was calculated using the BCVA worksheet, which was kept in the source data and the score was recorded in the eCRF.
  Between treatment comparison of 0.5 mg ranibizumab intravitreal injections driven by disease activity re-treatment criteria (Group II) versus 0.5 mg ranibizumab intravitreal injections driven by visual acuity stability criteria (Group I) based on the average BCVA change from Baseline to Month 1 through Month 12
Time Frame: From Baseline to Month 12
Population: FAS, modified LOCF for comparison between ranibizumab treatment groups.
Measure: Mean (Standard Deviation); unit: ETDRS letters
Arm/Group | Group I | Group II | Group III
Number analyzed (Participants) | 182 | 184 | 91
ETDRS letters
  Baseline: number analyzed (Participants) | 181 | 184 | 89
  Baseline | 53.7 (12.65) | 54.2 (13.01) | 52.6 (12.29)
  Average Month 1 to Month 12: number analyzed (Participants) | 181 | 184 | 89
  Average Month 1 to Month 12 | 64.8 (12.82) | 65.9 (13.26) | 61.2 (13.10)

4. Secondary Outcome: Mean Change From Baseline in Visual Acuity Over Time
Description: Best corrected visual acuity (BCVA) was tested using the ETDRS VA testing protocol. VA measurements were taken in a sitting position at an initial test distance of 4 meters using ETDRS charts. The overall BCVA score was calculated using the BCVA worksheet, which was kept in the source data and the score was recorded in the eCRF.
Time Frame: Change from baseline at months 3, 6, and 12
Population: FAS
Measure: Mean (Standard Deviation); unit: ETDRS letters
Arm/Group | Group I | Group II | Group III
Number analyzed (Participants) | 182 | 184 | 91
ETDRS letters
  Month 3: number analyzed (Participants) | 181 | 184 | 89
  Month 3 | 10.5 (9.13) | 10.8 (10.09) | 4.5 (9.35)
  Month 6: number analyzed (Participants) | 181 | 184 | 89
  Month 6 | 11.6 (10.66) | 12.1 (11.57) | 9.5 (10.50)
  Month 12: number analyzed (Participants) | 181 | 184 | 89
  Month 12 | 12.0 (11.50) | 13.1 (11.46) | 10.3 (12.69)

5. Secondary Outcome: Categorized BCVA Changes at Months 3, 6 and 12 Compared With Baseline for the Study Eye
Description: ETDRS VA testing protocol. VA measurements were taken in a sitting position at an initial test distance of 4 meters using ETDRS charts. The overall BCVA score was calculated using the BCVA worksheet, which was kept in the source data and the score was recorded in the eCRF.
Time Frame: From Baseline to Month 12
Population: FAS
Measure: Number; unit: Participants
Arm/Group | Group I | Group II | Group III
Number analyzed (Participants) | 182 | 184 | 91
Participants
  Gained≥15 letters or reached 84 letters-Month 3 | 58 | 59 | 15
  Gained≥10 letters or reached 84 letters-Month 3 | 97 | 107 | 24
  Gained≥15 letters or reached 84 letters-Month 6 | 71 | 73 | NA — Did not measure for this group as patients randomized to vPDT were allowed to receive ranibizumab from Month 3 onwards.
  Gained≥10 letters or reached 84 letters-Month 6 | 100 | 121 | NA — Did not measure for this group as patients randomized to vPDT were allowed to receive ranibizumab from Month 3 onwards.
  Gained≥15 letters or reached 84 letters-Month 12 | 81 | 75 | NA — Did not measure for this group as patients randomized to vPDT were allowed to receive ranibizumab from Month 3 onwards.
  Gained≥10 letters or reached 84 letters-Month 12 | 110 | 115 | NA — Did not measure for this group as patients randomized to vPDT were allowed to receive ranibizumab from Month 3 onwards.

6. Secondary Outcome: Mean Change From Baseline Over Time in Central Sub-field Thickness (CSFT)
Description: Central sub-field thickness (CSFT) is a variable assessed via Optical Coherence Tomography (OCT). OCT was performed prior to any study drug administration to assess presence of intra, subretinal fluid, or increase of CSFT.
Time Frame: Baseline, Month 3, Month 6, and Month 12
Measure: Mean (Standard Deviation); unit: micrometer
Arm/Group | Group I | Group II | Group III
Number analyzed (Participants) | 182 | 184 | 91
micrometer
  Month 3 | -66.4 (98.68) | -71.2 (81.28) | -29.1 (75.57)
  Month 6 | -70.7 (73.20) | -75.1 (80.90) | -59.3 (81.82)
  Month 12 | -79.4 (71.39) | -80.8 (85.93) | -66.0 (93.60)

7. Secondary Outcome: Number of Patients With CNV Leakage (Center Involvement) in the Study Eye at Baseline and Month 12
Description: CNV leakage is assessed via fluorescein angiography (center involvement) category: definite, questionable, absent, can't grade, and missing.
Time Frame: From Baseline until Month 12
Population: FAS
Measure: Number; unit: Participants
Arm/Group | Group I | Group II | Group III
Number analyzed (Participants) | 182 | 184 | 91
Participants
  Baseline - Definite | 164 | 160 | 76
  Baseline - Questionable | 1 | 3 | 0
  Baseline - Absent | 14 | 19 | 13
  Baseline - Can't Grade | 2 | 0 | 0
  Baseline - Missing | 1 | 2 | 2
  Month 12 - Definite | 34 | 43 | 26
  Month 12 - Questionable | 6 | 4 | 2
  Month 12 - Absent | 133 | 129 | 56
  Month 12 - Can't Grade | 2 | 2 | 0
  Month 12 - Missing | 7 | 6 | 7

8. Secondary Outcome: NEI-VFQ-25 - Change From Baseline to Month 3, 6 and 12
Description: The VFQ-25 consists of 25 vision related questions across 11 vision related subscales, including general vision, ocular pain, near activities, distance activities, social function, mental health, role difficulties, dependency, driving, color vision and peripheral vision, and a general health rating. Items are converted to a 0-100 scale on each subscale and for the composite score where higher scores represents better functioning.
Time Frame: Change from baseline at month 3, 6 and 12
Population: FAS
Measure: Mean (Standard Deviation); unit: Composite score
Arm/Group | Group I | Group II | Group III
Number analyzed (Participants) | 182 | 184 | 91
Composite score
  Month 3: number analyzed (Participants) | 175 | 179 | 89
  Month 3 | 4.7 (12.28) | 6.1 (13.49) | 1.7 (13.55)
  Month 6: number analyzed (Participants) | 176 | 180 | 89
  Month 6 | 5.0 (13.40) | 5.6 (15.42) | -0.1 (15.30)
  Month 12: number analyzed (Participants) | 177 | 180 | 89
  Month 12 | 4.4 (16.03) | 4.7 (16.92) | 1.3 (16.85)

9. Secondary Outcome: Number of Ranibizumab Injections Received in the Study Eye for the Ranibizumab Groups
Description: To assess treatment pattern with ranibizumab
Time Frame: From Baseline to Month 12
Population: Safety Set: all patients who received at least one application of study treatment & had at least one post-Baseline safety assessment. Patients were analyzed according to treatment received. One patient randomized to vPDT Group III received one ranibizumab injection prior to Month 3; this patient was analyzed under Group II in Safety Set
Measure: Mean (Standard Deviation); unit: Injections
Groups:
- Group III With 0.5mg Ranibizumab: verteporfin PDT with 0.5 mg ranibizumab from month 3
- Group III Without 0.5mg Ranibizumab: verteporfin PDT without 0.5 mg ranibizumab from month 3
Arm/Group | Group I | Group II | Group III With 0.5mg Ranibizumab | Group III Without 0.5mg Ranibizumab
Number analyzed (Participants) | 182 | 185 | 75 | 14
Injections
  Month 3 | 2.4 (0.53) | 2.1 (0.84) | NA (NA) — Did not measure for this group at month 3 | NA (NA) — Did not measure for this group at month 3
  Month 12 | 4.6 (2.44) | 3.9 (2.50) | 3.2 (2.25) | 3.8 (2.36)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Treatment, approximately 4 years.
Description: Analysis was done in the safety set: consisted of all patients who received at least one application of study treatment and had at least one post-Baseline safety assessment. Patients were analyzed according to treatment received. The statement that a patient had no AEs also constitutes a safety assessment.
  One patient randomized to vPDT Group III received one ranibizumab injection prior to Month 3; this patient was analyzed under Group II in Safety Set"
Groups:
- Group III With 0.5mg Ranibizumab: Visudyne PDT with 0.5mg ranibizumab from month 3
- Group III Without 0.5mg Ranibizumab: Visudyne PDT without 0.5mg ranibizumab from month 3
Arm/Group | Group I | Group II | Group III With 0.5mg Ranibizumab | Group III Without 0.5mg Ranibizumab
Serious Adverse Events (participants affected / at risk) | 7/182 | 15/185 | 8/75 | 0/14
Other Adverse Events (participants affected / at risk) | 102/182 | 116/185 | 50/75 | 8/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group I (N=182) | Group II (N=185) | Group III With 0.5mg Ranibizumab (N=75) | Group III Without 0.5mg Ranibizumab (N=14)
Arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 2 | 0 | 0
Retinal detachment (Fellow eye) (Eye disorders) | 0 | 1 | 1 | 0
Retinal detachment (Study eye) (Eye disorders) | 1 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Rectal polyp (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Varices oesophageal (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Endophthalmitis (Study eye) (Infections and infestations) | 0 | 0 | 1 | 0
Pharyngitis bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Physical examination abnormal (Investigations) | 0 | 0 | 1 | 0
Shock hypoglycaemic (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Oligoastrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0
Bladder hyperaemia (Renal and urinary disorders) | 0 | 1 | 0 | 0
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group I (N=182) | Group II (N=185) | Group III With 0.5mg Ranibizumab (N=75) | Group III Without 0.5mg Ranibizumab (N=14)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 1 | 0
Cataract (Study eye) (Eye disorders) | 2 | 1 | 0 | 0
Choroidal neovascularisation (Fellow eye) (Eye disorders) | 2 | 3 | 1 | 1
Choroidal neovascularisation (Study eye) (Eye disorders) | 1 | 2 | 0 | 0
Conjunctival deposit (Fellow eye) (Eye disorders) | 2 | 1 | 0 | 0
Conjunctival deposit (Study eye) (Eye disorders) | 2 | 1 | 0 | 0
Conjunctival haemorrhage (Study eye) (Eye disorders) | 8 | 14 | 2 | 0
Conjunctival hyperaemia (Study eye) (Eye disorders) | 2 | 1 | 0 | 0
Conjunctivitis allergic (Fellow eye) (Eye disorders) | 0 | 1 | 1 | 1
Conjunctivitis allergic (Study eye) (Eye disorders) | 1 | 2 | 1 | 1
Diplopia (Study eye) (Eye disorders) | 0 | 0 | 1 | 0
Dry eye (Fellow eye) (Eye disorders) | 2 | 2 | 0 | 1
Dry eye (Study eye) (Eye disorders) | 2 | 2 | 1 | 1
Exophthalmos (Fellow eye) (Eye disorders) | 3 | 0 | 0 | 0
Exophthalmos (Study eye) (Eye disorders) | 3 | 0 | 1 | 0
Eye pain (Fellow eye) (Eye disorders) | 4 | 3 | 0 | 0
Eye pain (Study eye) (Eye disorders) | 6 | 5 | 1 | 1
Eye pruritus (Study eye) (Eye disorders) | 2 | 2 | 0 | 1
Eye swelling (Fellow eye) (Eye disorders) | 0 | 1 | 0 | 1
Eye swelling (Study eye) (Eye disorders) | 3 | 1 | 1 | 1
Foreign body sensation in eyes (Study eye) (Eye disorders) | 0 | 0 | 1 | 0
Macular fibrosis (Study eye) (Eye disorders) | 1 | 2 | 1 | 0
Macular hole (Study eye) (Eye disorders) | 2 | 0 | 0 | 0
Metamorphopsia (Fellow eye) (Eye disorders) | 0 | 1 | 0 | 1
Metamorphopsia (Study eye) (Eye disorders) | 1 | 1 | 0 | 1
Ocular discomfort (Fellow eye) (Eye disorders) | 3 | 1 | 1 | 0
Ocular discomfort (Study eye) (Eye disorders) | 2 | 1 | 1 | 0
Ocular hypertension (Study eye) (Eye disorders) | 1 | 1 | 1 | 0
Pathologic myopia (Study eye) (Eye disorders) | 1 | 0 | 1 | 0
Photopsia (Study eye) (Eye disorders) | 0 | 1 | 1 | 0
Posterior capsule opacification (Study eye) (Eye disorders) | 2 | 1 | 0 | 0
Retinal haemorrhage (Fellow eye) (Eye disorders) | 2 | 4 | 0 | 2
Retinal haemorrhage (Study eye) (Eye disorders) | 2 | 2 | 1 | 1
Vision blurred (Study eye) (Eye disorders) | 0 | 6 | 0 | 0
Visual acuity reduced (Fellow eye) (Eye disorders) | 1 | 2 | 0 | 0
Visual acuity reduced (Study eye) (Eye disorders) | 2 | 0 | 2 | 0
Visual impairment (Study eye) (Eye disorders) | 2 | 0 | 0 | 0
Vitreous floaters (Study eye) (Eye disorders) | 0 | 0 | 1 | 0
Vitreous opacities (Fellow eye) (Eye disorders) | 0 | 2 | 0 | 0
Vitreous opacities (Study eye) (Eye disorders) | 1 | 2 | 0 | 0
Xerophthalmia (Fellow eye) (Eye disorders) | 6 | 7 | 1 | 0
Xerophthalmia (Study eye) (Eye disorders) | 7 | 7 | 2 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Glossitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Loose tooth (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 4 | 1 | 3 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 2 | 0 | 0 | 0
Peripheral swelling (General disorders) | 2 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 3 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 0 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 2 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 2 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 2 | 2 | 0
Allergy to chemicals (Immune system disorders) | 0 | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 1 | 0
Bronchitis (Infections and infestations) | 5 | 1 | 1 | 0
Conjunctivitis (Fellow eye) (Infections and infestations) | 1 | 6 | 3 | 1
Conjunctivitis (Study eye) (Infections and infestations) | 2 | 5 | 3 | 1
Cystitis (Infections and infestations) | 2 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 3 | 1 | 1 | 0
Gastroenteritis shigella (Infections and infestations) | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 3 | 1 | 0 | 0
Hordeolum (Study eye) (Infections and infestations) | 1 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 17 | 20 | 8 | 1
Periodontitis (Infections and infestations) | 2 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 2 | 3 | 0 | 0
Pulpitis dental (Infections and infestations) | 2 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 14 | 12 | 6 | 0
Urethritis (Infections and infestations) | 1 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 4 | 2 | 3 | 0
Vaginal infection (Infections and infestations) | 2 | 1 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 3 | 1 | 0 | 0
Spinal column injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 4 | 2 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 4 | 1 | 0 | 0
Bacterial test positive (Investigations) | 2 | 1 | 1 | 0
Blood glucose increased (Investigations) | 2 | 6 | 3 | 0
Blood pressure increased (Investigations) | 2 | 0 | 2 | 0
Blood uric acid increased (Investigations) | 7 | 2 | 1 | 0
Blood urine present (Investigations) | 1 | 1 | 2 | 0
Intraocular pressure increased (Fellow eye) (Investigations) | 2 | 4 | 1 | 0
Intraocular pressure increased (Study eye) (Investigations) | 2 | 4 | 1 | 0
Platelet count decreased (Investigations) | 1 | 0 | 1 | 0
Pregnancy test positive (Investigations) | 0 | 2 | 0 | 0
Protein urine present (Investigations) | 3 | 3 | 2 | 0
Red blood cells urine positive (Investigations) | 1 | 0 | 1 | 0
Urine ketone body present (Investigations) | 0 | 0 | 1 | 0
Urine leukocyte esterase positive (Investigations) | 2 | 0 | 0 | 0
Visual acuity tests abnormal (Study eye) (Investigations) | 3 | 3 | 3 | 0
White blood cell count decreased (Investigations) | 0 | 3 | 1 | 0
White blood cells urine positive (Investigations) | 1 | 1 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 3 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0
Rheumatic disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Diabetic neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 3 | 1 | 1 | 0
Facial neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 9 | 2 | 0
Migraine (Nervous system disorders) | 1 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 2 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 3 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 1 | 0
Breast hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 1 | 0
Breast swelling (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Menopausal symptoms (Reproductive system and breast disorders) | 1 | 0 | 1 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 1 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 10 | 5 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 2 | 0
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Arteriosclerosis (Vascular disorders) | 0 | 0 | 1 | 0
Diabetic vascular disorder (Vascular disorders) | 0 | 0 | 1 | 0
Hyperaemia (Study eye) (Vascular disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 7 | 2 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.